CLINICAL TRIAL: NCT06713785
Title: Personalised Electronic Record Supported Optimisation of Amlodipine for Patients With Hypertension
Acronym: PERSONAL HTN
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: 4.09.2020 decided to close the PERSONAL-HTN study without recruiting any patients because its approval by MHRA and HRA under CWoW coincided with the COVID-19 pandemic and lockdown in England
Sponsor: Queen Mary University of London (Other)
Collaborators: INNOVATEUK (Unknown); Closed Loop Medicine Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2019-11-14; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine

STUDY DESIGN:
Intervention Model Description: Single site, open label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amlodipine 0mg (Other): amlodipine dose 0mg Week 0 → 1mg Week 2 → 2mg Week 4 → 3mg Week 6 → 4mg Week 8 → 5mg Dose escalation to continue in 1mg increments to a maximum of 5mg
  Interventions: Drug: Amlodipine
- Amlodipine 5mg (Other): amlodipine dose 5mg Week 0 → 6mg Week 2 → 7mg Week 4 → 8mg Week 6 → 9mg Week 8 → 10mg Dose escalation to continue in 1mg increments to a maximum of 10mg
  Interventions: Drug: Amlodipine

INTERVENTIONS:
Drug: Amlodipine — Amlodipine 1mg/ml Oral Solution

SUMMARY:
The primary objective of the study is to assess precision dosing of amlodipine to deliver reductions in blood pressure in patients with primary hypertension and inadequate BP control by up-titration of amlodipine in 1mg increments

DETAILED DESCRIPTION:
Hypertension is the leading preventable cause of premature death worldwide. Globally, 1.39bn people are estimated to have hypertension, and it caused ≈10.7 million deaths in 2015. It is projected to affect more than 1.5 billion people around the world by 2025.

In the UK ~30% of adults have hypertension3; 9.5m have a diagnosis, and a further 5m people in England alone may have hypertension yet be unaware. The annual incidence of new cases is 5-8%5. Physician inertia (inadequate up-titration of treatment, especially from monotherapy) and poor patient adherence to treatment (especially when based on multiple pills) are now recognised as major factors contributing to poor BP control.

Amlodipine is a calcium-channel blocking drug which reduces blood pressure by relaxing blood vessels (especially veins) but this same effect makes it prone to causing fluid accumulation (oedema) in the lower limbs. Approved by the FDA in the United States in 1987, there is a large amount of evidence on its effectiveness and safety in reducing blood pressure and in treating stable angina. There appears to be a close relationship between wanted and unwanted effects. Finding the best dose of amlodipine for a patient could be useful in optimizing their blood pressure treatment. At present the tablet doses available are only 5mg and 10mg in the UK.

In the present study the investigators will investigate the relationship between patient beliefs about medicines using the Beliefs about Medicines Questionnaire (BMQ) developed by Horne, Weinman and Hankins (1999)13 and their adherence using the Morisky Medication Adherence Scale - 8 14. The investigators hypothesize that patients' tolerability of side effects (as measured by VAS) will be related to their beliefs about the necessity of medication (necessity concerns), their concerns about side effects and their adherence to medication.

This study will only look at doses within the current maximum licensed 10mg dose. The investigators will ask patients who have had previous problems with unwanted effects of amlodipine at conventional doses to have careful monitoring of blood pressure over 24 hours using an ambulatory blood pressure monitor. If blood pressure control on their maximum tolerated conventional dose of amlodipine (0 or 5mg) is inadequate (systolic daytime average =>135 mmHg and/or diastolic daytime average =>85 mmHg), then patients will be eligible for the study. Those taking 5mg amlodipine tablets daily will be given amlodipine liquid to take at the same 5mg dose to convert to liquid formulation dosing. Patients will be issued with standard home blood pressure monitors and will be asked to measure their blood pressure in the morning (three readings) before taking their tablet (trough treatment) and again in the evening (three readings). Patients will attend every two weeks, following screening with clinical history taking, haematology, biochemistry, HbA1c, routine physical examination and resting ECG. Every two weeks patients will have clinic blood pressure measurements and review of home BP monitoring

ELIGIBILITY:
Inclusion Criteria:

* - Age ≥18 years to 75 years
* Able to give consent
* Possession of a smart phone
* Confirmed diagnosis of hypertension by NICE/BIHS criteria on either 24h ABPM or repeated home measures of blood pressure, at any time.
* Previous experience of amlodipine and unwanted effects of the drug
* Willing to be re-challenged with amlodipine (if off treatment) or to try a higher dose than the 5mg currently treated with.
* Sub-optimal blood pressure control defined as daytime ABPM average systolic blood pressure of 135mmHg or greater, and/or daytime ABPM average diastolic blood pressure of 85mmHg or greater.
* Stable antihypertensive medication (ie. no dose adjustments, new Rx or stopped Rx in last 4 weeks for CCB, 8 weeks for diuretics, ACEi, ARB).
* Patients may be taking other blood pressure lowering medication, but these must be kept stable during assessment of eligibility and for the duration of the trial (except where essential to maintain patient safety).

Exclusion Criteria:

* - Unable to consent.
* Severe adverse reaction to amlodipine making re-challenge or dose increase unwise.
* Myocardial infarction, Acute Coronary Syndrome, stroke or Transient Ischaemic Attack in the 6 months prior to screening.
* Heart failure classed as NYHA class III or IV.
* Renal impairment with eGFR < 30ml/minute.
* Participation in another clinical trial, where the patient has received IMP in the last 3 months, except for MRC Aim-Hy with established medications and where patients can be screened after 6 weeks from final visit.
* Pregnant or lactating or female of childbearing potential not using adequate contraception

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-26 (Estimated); Primary Completion 2021-01-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
The difference in daytime ambulatory systolic blood pressure between baseline ABPM and post-titration ABPM on a personalized dose of amlodipine. | End of study 1 year
  pressure between baseline ABPM and post-titration ABPM on a personalized dose of amlodipine.

SECONDARY OUTCOMES:
Other clinically significant blood pressure measures which related to difference in measured blood pressure between baseline and EOS, especially AOBP clinic BP readings and home BP readings | End of study 1 year
  Other clinically significant blood pressure measures which related to difference in measured blood pressure between baseline and EOS, especially AOBP clinic BP readings and home BP readings
Feasibility of collecting data using a digital diary | End of study 1 year
  Feasibility of collecting data using a digital diary
Collect patient reported outcome data including satisfaction with medication regime using digital diary | Collect patient reported outcome data including satisfaction with medication regime using digital diary
  Collect patient reported outcome data including satisfaction with medication regime using digital diary
Patient feedback on the use of digital diary | End of study 1 year
  Patient feedback on the use of digital diary
Insight into number of patients achieving target BP of <135 and 85 at EOS | End of study 1 year
  Insight into number of patients achieving target BP of <135 and 85 at EOS
Insight into number of patients achieving reduction in systolic BP of ≥5mmHg at EOS | End of Study
  Insight into number of patients achieving reduction in systolic BP of ≥5mmHg at EOS
Insight into number of patients achieving reduction in systolic BP of ≥10mmHg EOS | EOS 1 year
  Insight into number of patients achieving reduction in systolic BP of ≥10mmHg EOS
Insight into number of patients achieving reduction in diastolic BP of ≥5mmHg at EOS | End of study 1 year
  Insight into number of patients achieving reduction in diastolic BP of ≥5mmHg at EOS

CONTACTS AND LOCATIONS:
Overall Officials: David Collier, Dr, Principal Investigator — Clinical Director

IPD SHARING:
Plan to Share IPD: Yes
Main study findings will be published on websites of the cardiovascular unit at Barts. Following primary publication of the trial results, fully anonymized trial data can be made available to interested researchers on request to the Chief Investigator.
  The sponsor retains the right to review all publications prior to submission or publication. Responsibility for ensuring accuracy of any publication from this study is delegated to the Chief Investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Post-trial, timeframe unspecified
Access Criteria: Approved authorised by CI and clinical/research team.